CLINICAL TRIAL: NCT00047762
Title: Open-Label, Multicenter, Dose-Escalation Study in Subjects w/Advanced Colorectal Cancer to Evaluate the Safety, Efficacy, and Pharmacokinetics of Tarceva in Combination w/5-Fluorouracil, Leucovorin, and Irinotecan and of Bevacizumab in Combination w/Tarceva, 5-Fluorouracil, Leucovorin, and Irinotecan
Brief Title: Safety, Efficacy, and Pharmacokinetics Study of Tarceva to Treat Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: OSI2520g
Record Dates: First submitted 2002-10-16; First posted 2002-10-18 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Erlotinib Hydrochloride; Bevacizumab

INTERVENTIONS:
Drug: Erlotinib (aka Tarceva or OSI-774)
Drug: Bevacizumab (aka Avastin or Rhu MAb VEGF)

SUMMARY:
The purpose of this study is test the safety of Tarceva, find the best dose, and see what effects (good and bad) it has on you and your colorectal cancer. The effects of Tarceva will be evaluated in combination with 5-fluorouracil, leucovorin, and irinotecan, with or without Bevacizumab.

ELIGIBILITY:
Subjects must fulfill all of the following criteria to be eligible for study entry:

* Signed informed consent
* At least 18 years of age
* Histologically confirmed metastatic colorectal adenocarcinoma of the colon or rectum

Resected or biopsied primary tumors or metastatic site will serve as the basis for histologic confirmation.

* Measurable disease (defined as at least one dimension >2 cm [>1 cm on spiral CT scans])
* ECOG performance status of 0 or 1
* Life expectancy >3 months
* Use of an effective means of contraception in men and in women of childbearing potential
* Ability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Indiana University Cancer Pavilion, Indianapolis, Indiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Mary Crowley Medical Research Center, Dallas, Texas